CLINICAL TRIAL: NCT00624195
Title: HIV Neurocognitive Disorders: A Randomized Clinical Trial of CNS-Targeted HAART
Brief Title: Clinical Trial of CNS-targeted HAART (CIT2)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ronald J Ellis, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 060154; R01MH058076-09A2 (NIH)
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: HIV Infections
Keywords: HIV Dementia; HAART; Cognitive Impairment; Antiretroviral Regimen; Viral Load; CNS Drug Penetration
MeSH Terms: conditions — HIV Infections; AIDS Dementia Complex; Cognitive Dysfunction | interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lamivudine, zidovudine drug combination; Emtricitabine; Lamivudine; abacavir, lamivudine drug combination; Zidovudine; abacavir, lamivudine, and zidovudine drug combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; abacavir; etravirine; Delavirdine; efavirenz; Nevirapine; amprenavir; tipranavir; Saquinavir; lopinavir-ritonavir drug combination; fosamprenavir; Ritonavir; Darunavir; Atazanavir Sulfate; Nelfinavir; Enfuvirtide; Maraviroc; Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CNS-targeted (Experimental): CNS-T will comprise two components: 1) initial selection of agents to optimize CNS penetration of the overall regimen; and 2) modification of the regimen if an interim pharmacokinetic (PK) assessment determines that plasma ARV exposure is not appropriate (overdosing, under dosing).
  Possible regimens include combinations of these FDA approved antiretroviral agents: Efavirenz/Emtricitabine/Tenofovir, Lamivudine/Zidovudine, Emtricitabine, Lamivudine, Abacavir/Lamivudine, Zidovudine, Abacavir/Lamivudine/Zidovudine, Emtricitabine/Tenofovir, Tenofovir, Abacavir, Etravirine, Delavirdine, Efavirenz, Nevirapine, Amprenavir, Tipranavir, Saquinavir, Lopinavir/ritonavir, Fosamprenavir, Ritonavir, Darunavir, Atazanavir, Nelfinavir, Enfuvirtide, Maraviroc, Raltegravir
  Interventions: Drug: FDA Approved Antiretroviral Therapy (see list below)
- non-CNS-targeted (Active Comparator): Subjects in the non-CNS-T (Comparison) arm will be randomized to receive a regimen (see list of FDA approved antiretrovirals listed below) designed to suppress plasma Viral Load, but not expected to have targeted CNS penetration.
  Combinations of FDA approved antiretroviral agents: Efavirenz/Emtricitabine/Tenofovir, Lamivudine/Zidovudine, Emtricitabine, Lamivudine, Abacavir/Lamivudine, Zidovudine, Abacavir/Lamivudine/Zidovudine, Emtricitabine/Tenofovir, Tenofovir, Abacavir, Etravirine, Delavirdine, Efavirenz, Nevirapine, Amprenavir, Tipranavir, Saquinavir, Lopinavir/ritonavir, Fosamprenavir, Ritonavir, Darunavir, Atazanavir, Nelfinavir, Enfuvirtide, Maraviroc, Raltegravir
  Interventions: Drug: FDA Approved Antiretroviral Therapy (see list below)

INTERVENTIONS:
Drug: FDA Approved Antiretroviral Therapy (see list below) — Combinations of FDA approved antiretroviral agents:
  Atripla, Combivir, Emtriva, Epivir, Epzicom, Retrovir, Trizivir, Truvada, Viread, Ziagen, Intelence, Rescriptor, Sustiva, Viramune, Agenerase, Aptivus, Invirase, Kaletra, Lexiva, Norvir, Prezista, Reyataz, Viracept, Fuzeon, Selzentry, Isentress
  Generic names: Efavirenz/Emtricitabine/Tenofovir, Lamivudine/Zidovudine, Emtricitabine, Lamivudine, Abacavir/Lamivudine, Zidovudine, Abacavir/Lamivudine/Zidovudine, Emtricitabine/Tenofovir, Tenofovir, Abacavir, Etravirine, Delavirdine, Efavirenz, Nevirapine, Amprenavir, Tipranavir, Saquinavir, Lopinavir/ritonavir, Fosamprenavir, Ritonavir, Darunavir, Atazanavir, Nelfinavir, Enfuvirtide, Maraviroc, Raltegravir
  Other Names: Atripla; Combivir; Emtriva; Epivir; Epzicom; Retrovir; Trizivir; Truvada; Viread; Ziagen; Intelence; Rescriptor; Sustiva; Viramune; Agenerase; Aptivus; Invirase; Kaletra; Lexiva; Norvir; Prezista; Reyataz; Viracept; Fuzeon; Selzentry; Isentress

SUMMARY:
CIT2 is a strategy for targeting HAART (Highly Active Antiretroviral Therapy) to the CNS (Central Nervous System) in patients with HIV associated neurocognitive impairment (HNCI).

The primary goal of this study is to evaluate the effectiveness of CNS-targeted (CNS-T) as compared to non-CNS-targeted (non-CNS-T) HAART in treating HNCI globally and in different domains of functioning known to be affected by HIV.

It is hypothesized that participants in the CNS-T arm will have greater improvement in neurocognitive functioning than those in the non-CNS-T arm.

The secondary goal of the study is to compare participants assigned to CNS-T and non-CNS-T HAART on measures of CNS and systemic HIV suppression (undetectable CSF and plasma VL).

It is also hypothesized that although CSF viral suppression will be more frequent in the CNS-T arm, plasma viral suppression will be similar in the two treatment arms.

DETAILED DESCRIPTION:
"HIV Neurocognitive Disorders: A Randomized Clinical Trial of CNS-targeted HAART" is a randomized, controlled clinical trial to assess the efficacy of a strategy for targeting highly active antiretroviral therapy (HAART) to the CNS in patients with HIV associated neurocognitive impairment (HNCI). Contemporary cohort studies have consistently demonstrated that HNCI remains a prevalent disorder in patients receiving HAART. HNCI is a significant burden to persons living with HIV infection, caregivers, and the healthcare system. Thus the development of effective treatment strategies is of critical public health importance.

This study is based on findings from a previous study. Briefly, among individuals with HNCI who initiated a new antiretroviral (ARV) therapy regimen, those receiving more highly CNS-penetrating ARV regimens were more likely to successfully suppress cerebrospinal fluid (CSF) viral load (VL), and those who achieved CSF suppression (VL < 50 c/mL) had better neurocognitive (NC) outcomes. These findings suggest that NC outcomes of ART may be enhanced by the planned application of an ARV selection and clinical monitoring strategy designed to optimize the treatment of CNS infection. In the future it will become increasingly important to consider CNS penetration issues in selecting ART regimens. The randomized clinical trial proposed here would provide the level of evidence needed to formulate ART guidelines specific to HNCI.

Subjects eligible for this trial will be individuals with HNCI who anticipate initiation of a new ARV regimen or substitution of their existing regimen following contemporary treatment guidelines. A total of 120 patients at 3 study sites will be randomized 1:1 to receive a CNS-targeted (CNS-T) ARV strategy versus a non-CNS-targeted (Comparison) strategy. The primary outcome, change in global neuropsychological (NP) performance, will be assessed at 16 weeks. CNS-T will comprise two components: 1) initial selection of agents to optimize CNS penetration of the overall regimen; and 2) modification of the regimen if an interim pharmacokinetic (PK) assessment determines that plasma ARV exposure is not appropriate (overdosing, underdosing).

ELIGIBILITY:
Inclusion Criteria:

* HIV infected- confirmed by ELISA or 2 prior viral loads >2000
* 18 years or older
* Under consideration to initiate or change their HAART regimens (based on current consensus treatment guidelines) as directed by their primary care physicians.
* Measurable HIV Neurocognitive Impairment (HNCI)
* Willing and able to undergo at least 3 lumbar punctures safely during the course of the study.
* Potential subjects must have a Karnofsky score of > or = to 60 within 60 days prior to study entry.
* Potential subjects must have a CD4 cell count obtained within 60 days prior to study entry.

Exclusion Criteria:

* Presence of serious illness, including HIV-related opportunistic infections, requiring systemic treatment and/or hospitalization until candidate either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 14 days prior to study entry.
* Presence of neurologic disorders other than HIV judged to be the principal cause of neurocognitive impairment.
* Presence of active, severe psychiatric disorders (e.g., major depression, schizophrenia) that would interfere with interpretation of the study evaluations or adherence to the study protocol or that might make their participation in the study problematic or unsafe.
* Presence of active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Use of any immunomodulator (interferons, interleukins, cyclosporine), vaccine, or investigational therapy including dexamethasone within 30 days prior to study entry.
* Inability to provide informed consent.
* Enrollment in other ARV treatment studies, unless the study is: 1) observational; 2) a compassionate use study that predated the current study; 3) one that does not require specific interventions (or one that does not dictate the regimen); or 4) one that does not include NP testing.
* A positive serum or urine pregnancy test, if female and of reproductive potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-03; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Ellis, MD, PhD, Principal Investigator — UCSD HIV Neurobehavioral Research Center
Locations (5):
- United States (5):
  - HIV Neurobehavioral Research Center, University of California San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins University- School of Medicine, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York

REFERENCES:
- [Background] May S, Letendre S, Haubrich R, McCutchan JA, Heaton R, Capparelli E, Ellis R. Meeting practical challenges of a trial involving a multitude of treatment regimens: an example of a multi-center randomized controlled clinical trial in neuroAIDS. J Neuroimmune Pharmacol. 2007 Mar;2(1):97-104. doi: 10.1007/s11481-006-9057-8. Epub 2007 Jan 10. PMID 18040832
- [Background] Letendre S, Marquie-Beck J, Capparelli E, Best B, Clifford D, Collier AC, Gelman BB, McArthur JC, McCutchan JA, Morgello S, Simpson D, Grant I, Ellis RJ; CHARTER Group. Validation of the CNS Penetration-Effectiveness rank for quantifying antiretroviral penetration into the central nervous system. Arch Neurol. 2008 Jan;65(1):65-70. doi: 10.1001/archneurol.2007.31. PMID 18195140
- [Result] Ellis RJ, Letendre S, Vaida F, Haubrich R, Heaton RK, Sacktor N, Clifford DB, Best BM, May S, Umlauf A, Cherner M, Sanders C, Ballard C, Simpson DM, Jay C, McCutchan JA. Randomized trial of central nervous system-targeted antiretrovirals for HIV-associated neurocognitive disorder. Clin Infect Dis. 2014 Apr;58(7):1015-22. doi: 10.1093/cid/cit921. Epub 2013 Dec 18. PMID 24352352
- See also: University of California, San Diego HIV Neurobehavioral Research Center Public Website — http://www.hnrc.ucsd.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-CNS-targeted: Subjects in the non-CNS-T (Comparison) arm will be randomized to receive a regimen designed to suppress plasma Viral Load, but not to expected to have targeted CNS penetration.
  Possible regimens include combinations of these FDA approved antiretroviral agents: Efavirenz/Emtricitabine/Tenofovir, Lamivudine/Zidovudine, Emtricitabine, Lamivudine, Abacavir/Lamivudine, Zidovudine, Abacavir/Lamivudine/Zidovudine, Emtricitabine/Tenofovir, Tenofovir, Abacavir, Etravirine, Delavirdine, Efavirenz, Nevirapine, Amprenavir, Tipranavir, Saquinavir, Lopinavir/ritonavir, Fosamprenavir, Ritonavir, Darunavir, Atazanavir, Nelfinavir, Enfuvirtide, Maraviroc, Raltegravir
Period: Overall Study
Arm/Group | CNS-targeted | Non-CNS-targeted
Started | 29 | 30
Completed | 26 | 23
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- CNS-targeted: CNS-T will comprise two components: 1) initial selection of agents to optimize CNS penetration of the overall regimen; and 2) modification of the regimen if an interim pharmacokinetic (PK) assessment determines that plasma ARV exposure is not appropriate (overdosing, underdosing).
- Non-CNS-targeted: Subjects in the non-CNS-T (Comparison) arm will be randomized to receive a regimen designed to suppress plasma Viral Load, but not to expected to have targeted CNS penetration.
- Total: Total of all reporting groups
Arm/Group | CNS-targeted | Non-CNS-targeted | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 30 | 59
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (8.8) | 43.6 (11.1) | 44.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychological Performance Change
Description: The outcome measure is change in performance from baseline to 16 weeks as measured by the global deficit score (GDS). The GDS is calculated by averaging the individual deficit scores from each neurocognitive test. Deficit scores for each test were calculated from age-, education-, gender-, and ethnicity-adjusted raw scores by methods that capture unexpectedly poor performance while ignoring better than expected performance. The GDS ranges in value from 0-5; higher scores indicate poorer cognitive functioning. Subjects with scores greater than or equal to 0.5 are considered cognitively impaired.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CNS-targeted | Non-CNS-targeted
Number analyzed (Participants) | 26 | 23
units on a scale | -0.27 (0.52) | -0.17 (0.41)

ADVERSE EVENTS:
Time Frame: Entry to 16 weeks
Arm/Group | CNS-targeted | Non-CNS-targeted
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/30
Other Adverse Events (participants affected / at risk) | 0/29 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNS-targeted (N=29) | Non-CNS-targeted (N=30)
Death (Infections and infestations) | 0 (0) | 1 (1)
Psychiatric Event (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNS-targeted (N=29) | Non-CNS-targeted (N=30)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No